CLINICAL TRIAL: NCT00716417
Title: A Phase Ib Open Label Study to Assess the Safety, Tolerability and Pharmacokinetics of Continuous Dosing With BIBW 2992 Combined With Two Different Regimens of Backbone Chemotherapy: Cisplatin Combined With 5 Fluorouracil and Cisplatin Combined With Paclitaxel in Patients With Advanced Solid Tumors.
Brief Title: Study to Determine the Maximum Tolerated Dose of BIBW 2992 (Afatinib) When Combined With Cisplatin/Paclitaxel or Cisplatin/5-FU in Patients With Advanced Solid Tumours
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: 1200.37; 2008-002613-43 (EudraCT Number: EudraCT)
Record Dates: First submitted 2008-07-15; First posted 2008-07-16 (Estimated); Results first posted 2013-10-16 (Estimated); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — Afatinib

ARMS (2):
- A. BIBW 2992-cisplatin-paclitaxel (Experimental): daily oral dose of BIBW 2992 combined with 3-weekly infusion of cisplatin-paclitaxel
  Interventions: Drug: BIBW 2992
- B. BIBW 2992-cisplatin-5FU (Experimental): daily oral dose of BIBW 2992 combined with 3-weekly infusion of cisplatin-5FU
  Interventions: Drug: BIBW 2992

INTERVENTIONS:
Drug: BIBW 2992 — In each arm, BIBW 2992 dose will be escalated to determine MTD. Starting dose will be 20mg daily followed by 40 mg (with the option of an intermediary dose of 30 mg) then 50mg daily. Dose escalation will stop at 50 mg. No intra patient dose escalation.
  Arms: B. BIBW 2992-cisplatin-5FU
Drug: BIBW 2992 — low to high dose, daily
  Arms: A. BIBW 2992-cisplatin-paclitaxel

SUMMARY:
Study to determine the maximum tolerated dose of BIBW 2992 when combined with backbone chemotherapies consisting in cisplatin plus paclitaxel or cisplatin plus 5 FU.

The overall safety, the pharmacokinetics and the anti-tumour efficacy will also be assessed.

ELIGIBILITY:
Inclusion criteria:

1. Patients with histologically or cytologically confirmed diagnosis of non resectable and / or metastatic cancer, preferably squamous cell carcinomas of head and neck, oesophagus, lung or cervix
2. Indication for a standard treatment with either cisplatin plus paclitaxel or cisplatin plus 5 FU as judged by the investigator
3. Age 18 years or older.
4. Life expectancy of at least three (3) months.
5. Written informed consent that is consistent with ICH-GCP guidelines.
6. Eastern Cooperative Oncology Group (ECOG) performance score less or equal 2.
7. Patients must have recovered from any therapy-related toxicity from previous chemo-, hormone-, immuno-, or radiotherapies.
8. Patients recovered from previous surgery.

Exclusion criteria:

1. Active infectious disease.
2. Gastrointestinal disorders that may interfere with the absorption of the study drug or chronic diarrhoea.
3. Serious illness or concomitant non-oncological disease considered by the investigator to be incompatible with the protocol.
4. Patients with untreated or symptomatic brain metastases. Patients with treated, asymptomatic brain metastases are eligible if there has been no change in brain disease status for at least four (4) weeks, no history of cerebral oedema or bleeding in the past four (4) weeks and no requirement for steroids or anti-epileptic therapy.
5. Cardiac left ventricular function with resting ejection fraction less than 50%
6. Absolute neutrophil count (ANC) less than 1500 / mm3.
7. Platelets count less than 100 000/mm3.
8. Bilirubin more than 1.5 x upper limit of institutional norm.
9. Aspartate amino transferase (AST) or alanine amino transferase (ALT) more than 3 x upper limit of institutional norm.
10. Serum creatinine more than 1.5 x upper limit of institutional norm.
11. Women and men sexually active and unwilling to use a medically acceptable method of contraception.
12. Pregnancy or breast-feeding.
13. Treatment with other investigational drugs; chemotherapy, immunotherapy, or radiotherapy or participation in another clinical study with anti-cancer therapy within the past 4 weeks before start of therapy or concomitantly with this study.
14. Treatment with an EGFR- or HER2 inhibiting drug within the past four weeks before start of therapy or concomitantly with this study (2 weeks for trastuzumab).
15. Patients unable to comply with the protocol.
16. Active alcohol or drug abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2008-07-01 (Actual); Primary Completion 2010-07-01 (Actual); Study Completion 2010-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (3):
- Belgium (3):
  - 1200.37.3202 Boehringer Ingelheim Investigational Site, Brussels
  - 1200.37.3201 Boehringer Ingelheim Investigational Site, Edegem
  - 1200.37.3203 Boehringer Ingelheim Investigational Site, Ghent

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section "Time Frame" are fulfilled, researchers can use the following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: One year after the approval has been granted by major Regulatory Authorities and after the primary manuscript has been accepted for publication, or after termination of the development program.
Access Criteria: For study documents - upon signing of a "Document Sharing Agreement". For study data - 1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.mystudywindow.com/msw/datasharing

RESULTS

PARTICIPANT FLOW:
Groups:
- Pac175 + Cis50 + Afatinib20: Patients received continous daily dosing with Afatinib 20mg film-coated tablets over 21 day treatment cycles and infusions of Paclitaxel 175mg/m^2 and Cisplatin 50mg/m^2 on day 1 of each cycle. Treatment until disease progression or toxicity.
- Pac175 + Cis75 + Afatinib20: Patients received continous daily dosing with Afatinib 20mg film-coated tablets over 21 day treatment cycles and infusions of Paclitaxel 175mg/m^2 and Cisplatin 75mg/m^2 on day 1 of each cycle. Treatment until disease progression or toxicity.
- Pac175 + Cis75 + Afatinib30: Patients received continous daily dosing with Afatinib 30mg film-coated tablets over 21 day treatment cycles and infusions of Paclitaxel 175mg/m^2 and Cisplatin 75mg/m^2 on day 1 of each cycle. Treatment until disease progression or toxicity.
- Pac175 + Cis75 + Afatinib40: Patients received continous daily dosing with Afatinib 40mg film-coated tablets over 21 day treatment cycles and infusions of Paclitaxel 175mg/m^2 and Cisplatin 75mg/m^2 on day 1 of each cycle. Treatment until disease progression or toxicity.
- Pac175 + Cis75 + Afatinib50: Patients received continous daily dosing with Afatinib 50mg film-coated tablets over 21 day treatment cycles and infusions of Paclitaxel 175mg/m^2 and Cisplatin 75mg/m^2 on day 1 of each cycle. Treatment until disease progression or toxicity.
- Cis75 + 5FU750 + Afatinib20: Patients received continous daily dosing with Afatinib 20mg film-coated tablets over 21 day treatment cycles and infusions of 5-Fluorouracil 750mg/m^2 and Cisplatin 75mg/m^2 on day 1 of each cycle. Treatment until disease progression or toxicity.
- Cis75 + 5FU750 + Afatinib30: Patients received continous daily dosing with Afatinib 30mg film-coated tablets over 21 day treatment cycles and infusions of 5-Fluorouracil 750mg/m^2 and Cisplatin 75mg/m^2 on day 1 of each cycle. Treatment until disease progression or toxicity.
- Cis75 + 5FU750 + Afatinib40: Patients received continous daily dosing with Afatinib 40mg film-coated tablets over 21 day treatment cycles and infusions of 5-Fluorouracil 750mg/m^2 and Cisplatin 75mg/m^2 on day 1 of each cycle. Treatment until disease progression or toxicity.
- Cis100 + 5FU750 + Afatinib30: Patients received continous daily dosing with Afatinib 30mg film-coated tablets over 21 day treatment cycles and infusions of 5-Fluorouracil 750mg/m^2 and Cisplatin 100mg/m^2 on day 1 of each cycle. Treatment until disease progression or toxicity.
- Cis100 + 5FU1000 + Afatinib30: Patients received continous daily dosing with Afatinib 30mg film-coated tablets over 21 day treatment cycles and infusions of 5-Fluorouracil 1000mg/m^2 and Cisplatin 100mg/m^2 on day 1 of each cycle. Treatment until disease progression or toxicity.
Period: Overall Study
Arm/Group | Pac175 + Cis50 + Afatinib20 | Pac175 + Cis75 + Afatinib20 | Pac175 + Cis75 + Afatinib30 | Pac175 + Cis75 + Afatinib40 | Pac175 + Cis75 + Afatinib50 | Cis75 + 5FU750 + Afatinib20 | Cis75 + 5FU750 + Afatinib30 | Cis75 + 5FU750 + Afatinib40 | Cis100 + 5FU750 + Afatinib30 | Cis100 + 5FU1000 + Afatinib30
Started | 3 | 6 | 5 | 11 | 1 | 3 | 7 | 3 | 5 | 3
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 6 | 5 | 11 | 1 | 3 | 7 | 3 | 5 | 3
Not completed — Adverse Event | 0 | 0 | 2 | 1 | 0 | 0 | 3 | 1 | 0 | 3
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Progressive disease | 3 | 5 | 3 | 8 | 0 | 3 | 3 | 1 | 5 | 0
Not completed — Dose limiting toxicity (DLT) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — On patient request due to toxicities | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pac175 + Cis50 + Afatinib20 | Pac175 + Cis75 + Afatinib20 | Pac175 + Cis75 + Afatinib30 | Pac175 + Cis75 + Afatinib40 | Pac175 + Cis75 + Afatinib50 | Cis75 + 5FU750 + Afatinib20 | Cis75 + 5FU750 + Afatinib30 | Cis75 + 5FU750 + Afatinib40 | Cis100 + 5FU750 + Afatinib30 | Cis100 + 5FU1000 + Afatinib30 | Total
Number analyzed (Participants) | 3 | 6 | 5 | 11 | 1 | 3 | 7 | 3 | 5 | 3 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.7 (14.0) | 61.8 (15.6) | 61.8 (5.9) | 58.1 (7.8) | 54.0 (NA) — only one patient in this group | 52.7 (9.7) | 53.1 (16.1) | 65.0 (8.5) | 59.2 (14.4) | 63.7 (9.3) | 58.58 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 2 | 3 | 0 | 0 | 2 | 2 | 3 | 1 | 19
  Male | 0 | 3 | 3 | 8 | 1 | 3 | 5 | 1 | 2 | 2 | 28

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLT) in the First Cycle for the Determination of the Maximum Tolerated Dose (MTD)
Description: Number of participants with DLT in the first cycle (21 days) for the determination of the MTD.
Time Frame: 21 days
Population: Treated Set (TS) - TS consisted of all patients who were dispensed study medication and have taken at least 1 dose of Afatinib.
Measure: Number; unit: Participants
Arm/Group | Pac175 + Cis50 + Afatinib20 | Pac175 + Cis75 + Afatinib20 | Pac175 + Cis75 + Afatinib30 | Pac175 + Cis75 + Afatinib40 | Pac175 + Cis75 + Afatinib50 | Cis75 + 5FU750 + Afatinib20 | Cis75 + 5FU750 + Afatinib30 | Cis75 + 5FU750 + Afatinib40 | Cis100 + 5FU750 + Afatinib30 | Cis100 + 5FU1000 + Afatinib30
Number analyzed (Participants) | 3 | 6 | 5 | 11 | 1 | 3 | 7 | 3 | 5 | 3
Participants | 0 | 0 | 2 | 2 | 1 | 0 | 0 | 2 | 0 | 2

2. Primary Outcome: Maximum Tolerated Dose (MTD) for Regimen A and Regimen B
Description: The MTD was determined using a standard 3 +3 dose escalation cohort design. The sample size and the number of patients who receive each dose in this design depends on the frequency of DLT at each dose level in cycle 1.
Time Frame: 21 days
Population: as for outcome 1
Measure: Number; unit: mg/m^2
Groups:
- Pac + Cis + Afatinib (Regimen A): Patients received continous daily dosing with Afatinib film-coated tablets over 21 day treatment cycles and infusions of Paclitaxel and Cisplatin on day 1 of each cycle in 5 dose levels as outlined in first primary endpoint.
- 5FU + Cis + Afatinib (Regimen B): Patients received continous daily dosing with Afatinib film-coated tablets over 21 day treatment cycles and infusions of 5-Fluorouracil and Cisplatin on day 1 of each cycle in 5 dose levels as outlined in first primary endpoint.
Arm/Group | Pac + Cis + Afatinib (Regimen A) | 5FU + Cis + Afatinib (Regimen B)
Number analyzed (Participants) | 26 | 21
mg/m^2
  Maximum tolerated dose - Afatinib | 20 | 30
  Maximum tolerated dose - Cisplatin | 75 | 100
  Maximum tolerated dose - Pac (A) or 5-FU (B) | 175 | 750

3. Secondary Outcome: Number of Patients With Objective Response
Description: Objective tumor response based on response evaluation criteria in solid tumors (RECIST) version 1.0. Objective response is defined as complete response (CR) and partial response (PR).
Time Frame: Tumor assessment were performed at screening and every 2nd cycle until end of follow up (=end of treatment + 30 days +/- 7 days)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Pac175 + Cis50 + Afatinib20 | Pac175 + Cis75 + Afatinib20 | Pac175 + Cis75 + Afatinib30 | Pac175 + Cis75 + Afatinib40 | Pac175 + Cis75 + Afatinib50 | Cis75 + 5FU750 + Afatinib20 | Cis75 + 5FU750 + Afatinib30 | Cis75 + 5FU750 + Afatinib40 | Cis100 + 5FU750 + Afatinib30 | Cis100 + 5FU1000 + Afatinib30
Number analyzed (Participants) | 3 | 6 | 5 | 11 | 1 | 3 | 7 | 3 | 5 | 3
Participants | 1 | 0 | 0 | 4 | 0 | 1 | 0 | 0 | 0 | 0

4. Secondary Outcome: Maximum Concentration of Afatinib in Plasma at Steady State (Cmax,ss)
Description: Cmax,ss represents the maximum concentration of afatinib in plasma at steady state
Time Frame: 0.05hours (h) before administration and 1h, 2h, 2h 55 minutes (min), 4h, 4h 30min, 5h, 6h, 8h, 10h, 24h, 48h, 216h, 480h after administration
Population: The pharmacokinetic analysis set includes all patients who took at least one dose of trial medication and provided at least one blood sample following drug administration. Values were excluded from descriptive statistics when a comparison with plasma concentrations in the same treatment group was impossible.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Pac175 + Cis50 + Afatinib20 | Pac175 + Cis75 + Afatinib20 | Pac175 + Cis75 + Afatinib30 | Pac175 + Cis75 + Afatinib40 | Pac175 + Cis75 + Afatinib50 | Cis75 + 5FU750 + Afatinib20 | Cis75 + 5FU750 + Afatinib30 | Cis75 + 5FU750 + Afatinib40 | Cis100 + 5FU750 + Afatinib30 | Cis100 + 5FU1000 + Afatinib30
Number analyzed (Participants) | 3 | 4 | 2 | 4 | 0 | 3 | 6 | 1 | 3 | 1
ng/mL | 22.1 (22.5) | 18.0 (24.9) | 17.7 (13.2) | 32.1 (79.2) |  | 48.9 (26.0) | 57.0 (41.1) | 32.7 (NA) — Not calculable. If N= 1 individual values are displayed. | 13.4 (28.9) | 17.3 (NA) — Not calculable. If N= 1 individual values are displayed.

ADVERSE EVENTS:
Time Frame: First administration of trial medication until 28 days after last administration of trial medication
Arm/Group | Pac175 + Cis50 + Afatinib20 | Pac175 + Cis75 + Afatinib20 | Pac175 + Cis75 + Afatinib30 | Pac175 + Cis75 + Afatinib40 | Pac175 + Cis75 + Afatinib50 | Cis75 + 5FU750 + Afatinib20 | Cis75 + 5FU750 + Afatinib30 | Cis75 + 5FU750 + Afatinib40 | Cis100 + 5FU750 + Afatinib30 | Cis100 + 5FU1000 + Afatinib30
Serious Adverse Events (participants affected / at risk) | 1/3 | 5/6 | 4/5 | 7/11 | 1/1 | 2/3 | 6/7 | 3/3 | 1/5 | 3/3
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 5/5 | 11/11 | 1/1 | 3/3 | 7/7 | 3/3 | 5/5 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pac175 + Cis50 + Afatinib20 (N=3) | Pac175 + Cis75 + Afatinib20 (N=6) | Pac175 + Cis75 + Afatinib30 (N=5) | Pac175 + Cis75 + Afatinib40 (N=11) | Pac175 + Cis75 + Afatinib50 (N=1) | Cis75 + 5FU750 + Afatinib20 (N=3) | Cis75 + 5FU750 + Afatinib30 (N=7) | Cis75 + 5FU750 + Afatinib40 (N=3) | Cis100 + 5FU750 + Afatinib30 (N=5) | Cis100 + 5FU1000 + Afatinib30 (N=3)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 3 | 4 | 0 | 1 | 1 | 3 | 0 | 0
Duodenal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 2 | 2 | 0 | 1 | 2 | 2 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 0 | 1 | 3 | 1 | 1 | 1
Asthenia (General disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1
General physical health deterioration (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Brain abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 2 | 2 | 2 | 1 | 3
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 1
Food intolerance (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 1 | 3 | 0 | 0 | 0 | 1 | 0 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pac175 + Cis50 + Afatinib20 (N=3) | Pac175 + Cis75 + Afatinib20 (N=6) | Pac175 + Cis75 + Afatinib30 (N=5) | Pac175 + Cis75 + Afatinib40 (N=11) | Pac175 + Cis75 + Afatinib50 (N=1) | Cis75 + 5FU750 + Afatinib20 (N=3) | Cis75 + 5FU750 + Afatinib30 (N=7) | Cis75 + 5FU750 + Afatinib40 (N=3) | Cis100 + 5FU750 + Afatinib30 (N=5) | Cis100 + 5FU1000 + Afatinib30 (N=3)
Anaemia (Blood and lymphatic system disorders) | 2 | 4 | 1 | 6 | 0 | 1 | 3 | 2 | 2 | 2
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 3 | 0 | 6 | 0 | 2 | 1 | 1 | 2 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 2 | 1 | 1 | 2
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bundle branch block right (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Conduction disorder (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Deafness (Ear and labyrinth disorders) | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0
Deafness unilateral (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 2 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dry eye (Eye disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye irritation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eye swelling (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Visual acuity reduced (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 2 | 4 | 0 | 2 | 1 | 1 | 1 | 0
Anorectal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 2 | 1 | 2 | 0 | 2 | 2 | 1 | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 2 | 2 | 6 | 1 | 2 | 5 | 0 | 3 | 3
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 2 | 1 | 0 | 0 | 2 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lip disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lip dry (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 4 | 3 | 8 | 0 | 2 | 5 | 1 | 2 | 3
Oral pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 1 | 0 | 2 | 0 | 1 | 1 | 1 | 2 | 1
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1 | 4 | 2 | 1 | 0 | 1 | 1 | 3 | 2
Asthenia (General disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Catheter site pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 2 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 2 | 2 | 0 | 10 | 0 | 1 | 6 | 2 | 3 | 2
Feeling cold (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Localised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 1
Oedema (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 2 | 0 | 1 | 0 | 0 | 1 | 1 | 3 | 0
Pain (General disorders) | 1 | 0 | 2 | 1 | 0 | 1 | 2 | 0 | 1 | 0
Pyrexia (General disorders) | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 2 | 0 | 1
Hepatic pain (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Cystitis (Infections and infestations) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Eye infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Furuncle (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Genital infection fungal (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Klebsiella infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nail infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Omphalitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oral fungal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1
Urinary tract infection enterococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract infection fungal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vaginal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Medication error (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Blood alkaline phosphatase (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 2 | 2
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood phosphorus decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood urea increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ejection fraction decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Electrocardiogram ST segment depression (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Electrocardiogram ST segment elevation (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Glomerular filtration rate decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 1
White blood cell count increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 3 | 2 | 4 | 0 | 0 | 2 | 1 | 3 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fluid imbalance (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 3 | 0 | 1 | 3 | 3 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 2 | 2 | 6 | 0 | 0 | 2 | 0 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypercreatinaemia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 2 | 0 | 1 | 0 | 1 | 1 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ageusia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 3 | 1 | 2 | 0 | 1 | 0 | 1 | 2 | 2
Dysgeusia (Nervous system disorders) | 0 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 1 | 1
Headache (Nervous system disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Neurotoxicity (Nervous system disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Sensory loss (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 2 | 2 | 2 | 0 | 0 | 1 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depressed mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 2 | 4 | 0 | 0 | 1 | 0 | 0 | 0
Self esteem inflated (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oliguria (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Stress urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Testicular swelling (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 2 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 2 | 0 | 1 | 3 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 3 | 0 | 1 | 1 | 1 | 2 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 2 | 0 | 1 | 2 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 2 | 2 | 4 | 0 | 0 | 1 | 1 | 2 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nail pitting (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 2 | 0 | 5 | 0 | 2 | 1 | 1 | 1 | 1
Skin fissures (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1
Skin fragility (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 2 | 1
Hypotension (Vascular disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Venous thrombosis limb (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication